CLINICAL TRIAL: NCT00796562
Title: A Phase II Trial of Myeloablative Conditioning and Transplantation of Partially HLA-mismatched Bone Marrow for Patients With Hematologic Malignancies
Brief Title: Safety Study of Bone Marrow Transplant Using Mismatched Tissue Followed by Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0820; NA_00015795 (Other: JHMIRB); KL2RR025006 (NIH)
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: MDS; Leukemias; Lymphomas
Keywords: Leukemia; Lymphoma; Hematologic malignancies; ALL; AML; MDS; Transplantation; Mismatched; Haploidentical; Busulfan; Cyclophosphamide; Cellcept; Tacrolimus; TBI; CMMOL; CML; JMML
MeSH Terms: conditions — Leukemia; Lymphoma; Hematologic Neoplasms | interventions — Busulfan; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Myeloablative haploidentical BMT (Experimental): * All participants except those with acute lymphoblastic leukemia and lymphoblastic lymphoma: Busulfan will be administered 1 mg/kg oral (or 0.8 mg/kg IV) four times per day for four days, followed by cyclophosphamide 50 mg/kg once per day for two days.
  * Participants with acute lymphocytic leukemia or lymphoblastic lymphoma: Cyclophosphamide will be administered 50 mg/kg once per day for two days, followed by total body irradiation at 300 cGy per day for four days.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Radiation: Total body irradiation

INTERVENTIONS:
Drug: Busulfan — Participant will receive Busulfan injections, 4 times a day for 4 days with dilantin prophylaxis (in patients 10 years of age or older). Busulfan levels in the blood will be measured and dose adjusted, if needed.
Drug: Cyclophosphamide — Patient will receive Cy by IV once a day for 2 days.
  Other Names: Cy; Cytoxan; CTX
Radiation: Total body irradiation — Patients will receive TBI once a day for 4 days.
  Other Names: TBI

SUMMARY:
The purpose of this study is to see if giving high dose chemotherapy and total body irradiation before and repeating high dose chemotherapy after a bone marrow transplant could reduce the incidence of graft rejection and disease for patients with blood cancers

DETAILED DESCRIPTION:
Allogeneic blood or marrow transplantation (alloBMT), following either marrow-ablative or nonmyeloablative conditioning, is a potentially curative treatment for a variety of hematologic malignancies and non-malignant hematologic disorders. Of all the potential sources of allografts, transplantation of stem cells from a human leukocyte antigen (HLA)-matched sibling has generally produced the best overall outcomes, i.e. overall and progression-free survival. Unfortunately, only about a third of candidates for alloBMT have HLA-matched siblings.

For patients who lack HLA-matched siblings, there are three alternative sources of stem cells for alloBMT: 1) volunteer unrelated donors; 2) umbilical cord blood; and 3) partially HLA-mismatched, or haploidentical, related donors. Since any patient shares exactly one HLA haplotype with each biological parent or child and half of siblings, an eligible haploidentical donor can be identified rapidly in nearly all cases. However, haploidentical BMT has been associated with significant risks of graft rejection and severe GVHD, which are manifestations of excessive alloreactivity by host and donor T cells, respectively.

The risk of severe GVHD may be reduced in intensively conditioned recipients of grafts that have been rigorously depleted of mature T cells or selectively depleted of alloreactive T cells, but the risks of serious infection and death from prolonged immune compromise in these patients remains high. Cyclophosphamide(Cy) is a highly immunosuppressive antineoplastic agent that has an established role in conditioning for alloBMT.

Typically, the drug is administered prior to transplantation to prevent graft rejection by suppressing the host immune system. However, pre-transplantation conditioning with Cy increases the risk of GVHD following allogeneic T cell infusion in mouse models. In contrast, administration of a properly timed, high dose of Cy after BMT inhibits both graft rejection and GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphocytic leukemia in high risk CR1
* Acute myeloid leukemia in CR1
* Therapy-related AML
* RAEB with >5% and <20% bone marrow blasts
* Chronic myelogenous leukemia beyond 1st chronic phase; Patients cannot be in blast crisis
* CMMoL
* JMML
* Chemotherapy-resistant Hodgkins Lymphoma or intermediate or high grade Non-Hodgkins lymphoma (Less than a PR after standard or salvage chemotherapy)
* Mantle cell lymphoma: chemotherapy refractory (Less than a PR after standard or salvage chemotherapy) or patients beyond CR1 with chemosensitive disease
* Follicular Lymphoma, Grade 3
* Transformed indolent lymphomas

Exclusion Criteria:

* Poor cardiac function: left ventricular ejection fraction <45% as determined by MUGA or ECHO. For pediatric patients LVEF <45% or a shortening fraction below normal limits for age.
* Poor pulmonary function: FEV1 and FVC <50% predicted for patients who have not received thoracic or mantle irradiation. For patients who have received thoracic or mantle irradiation, FEV1 and FVC <70% predicted or DLCO < 50 of predicted. For children unable to perform PFTs because of developmental stage pulse oximetry < 85% on RA
* Poor liver function: bilirubin >2 mg/dl (not due to hemolysis, Gilbert's or primary malignancy)
* Poor renal function: Creatinine >2.0mg/dl or creatinine clearance
* HIV-positive
* Positive leukocytotoxic crossmatch
* Women of childbearing potential who currently are pregnant or who are not practicing adequate contraception
* Uncontrolled viral, bacterial, or fungal infections Patients with symptoms consistent with RSV, influenza A, B, or parainfluenza at the time of enrollment will be assayed for the above viruses and if positive are not eligible for the trial until they are no longer symptomatic (patients may have continued assay positivity for a period of time post resolution of symptoms secondary to the nature of the assay.
* Indolent lymphomas (Follicular Grade 1 and 2, marginal zone, chronic lymphocytic leukemia, small lymphocytic lymphoma, MALT)

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Symons, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fine J.P. and Gray, R.J. (1999), A proportional hazards model for the subdistribution of a competing risk, Journal of the American Statistical Association, 94:496-509.
- [Derived] Symons HJ, Zahurak M, Cao Y, Chen A, Cooke K, Gamper C, Klein O, Llosa N, Zambidis ET, Ambinder R, Bolanos-Meade J, Borrello I, Brodsky R, DeZern A, Gojo I, Showel M, Swinnen L, Smith BD, Luznik L, Jones RJ, Fuchs EJ. Myeloablative haploidentical BMT with posttransplant cyclophosphamide for hematologic malignancies in children and adults. Blood Adv. 2020 Aug 25;4(16):3913-3925. doi: 10.1182/bloodadvances.2020001648. PMID 32813874

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants were screen failures.
Period: Overall Study
Arm/Group | Myeloablative Haploidentical BMT
Started | 96
Completed | 47
Not Completed | 49
Not completed — Death | 49

BASELINE CHARACTERISTICS:
Population: The entire set of participants was analyzed as one group, and the analysis was planned this way from the beginning of the study.
Arm/Group | Myeloablative Haploidentical BMT
Number analyzed (Participants) | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 80
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 42 [1 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Engraftment as Measured by Donor Chimerism
Description: Percentage of participants who achieved donor chimerism >=95%.
Time Frame: Day 60
Population: 8 participants were not evaluable for this outcome because they died prior to Day 60.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Haploidentical BMT
Number analyzed (Participants) | 88
percentage of participants | 91 [83 to 96]

2. Secondary Outcome: Non-relapse Mortality
Description: Number of participants deceased for reasons other than disease relapse or progression.
Time Frame: Day 100, 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Haploidentical BMT
Number analyzed (Participants) | 96
Participants
  100 days | 10
  1 year | 10

3. Secondary Outcome: Acute GVHD
Description: Percentage of participants who experience grade II-IV or III-IV acute graft-versus-host-disease (GVHD) by Przepiorka criteria. The stages are defined as follows:
  * Stage II: Rash on >50% of skin, bilirubin 2-3 mg/dL, or diarrhea 500-1000 mL/day
  * Stage III: Bilirubin 3-15 mg/dL or diarrhea >1000 mL/day
  * Stage IV: Generalized erythroderma with bullae or bilirubin >15 mg/dL This outcome was estimated using proportional subdistribution hazard regression model for competing risks (Fine and Gray 1999)
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Haploidentical BMT
Number analyzed (Participants) | 96
percentage of participants
  Grade II-IV | 11 [5 to 18]
  Grade III-IV | 4 [0 to 8]

4. Secondary Outcome: Chronic GVHD
Description: Percentage of participants who experience chronic GVHD. Chronic GVHD is graded using NIH consensus criteria and Seattle criteria. This outcome was estimated using proportional subdistribution hazard regression model for competing risks (Fine and Gray 1999)
Time Frame: 6 months, 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Haploidentical BMT
Number analyzed (Participants) | 96
percentage of participants
  6 months | 4 [0 to 8]
  12 months | 15 [8 to 22]

5. Secondary Outcome: Survival
Description: Percentage of participants alive (overall survival) and alive without disease relapse, progression, or diagnosis of myeloid malignancy (event-free survival). Estimated using Kaplan-Meier method.
Time Frame: 1 year, 2 years, 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Haploidentical BMT
Number analyzed (Participants) | 96
percentage of participants
  Overall survival, 1 year | 73 [65 to 82]
  Overall survival, 2 years | 57 [48 to 68]
  Overall survival, 3 years | 54 [44 to 65]
  Event-free survival, 1 year | 58 [48 to 69]
  Event-free survival, 2 years | 52 [42 to 63]
  Event-free survival, 3 years | 50 [41 to 62]

6. Secondary Outcome: Relapse
Description: Percentage of participants who experienced disease progression or relapse. This outcome was estimated using proportional subdistribution hazard regression model for competing risks (Fine and Gray 1999)
Time Frame: 1 year, 3 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Haploidentical BMT
Number analyzed (Participants) | 96
percentage of participants
  1 year | 35 [26 to 45]
  3 years | 43 [33 to 553]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Only the following adverse events were collected per protocol: non-relapse mortality in the first 100 days after BMT; graft failure; and all unexpected events considered significant by the principal investigator. Adverse events were assessed weekly through Day 60 and at Days 180, 365, and 730.
Arm/Group | Myeloablative Haploidentical BMT
All-Cause Mortality (participants affected / at risk) | 49/96
Serious Adverse Events (participants affected / at risk) | 22/96
Other Adverse Events (participants affected / at risk) | 37/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative Haploidentical BMT (N=96)
Altered mental status (Nervous system disorders) | 1 (1)
Aspergillosis (Infections and infestations) | 1 (1)
BK virus (Infections and infestations) | 2 (2)
Bleeding (General disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Cytomegalovirus (Infections and infestations) | 1 (1)
Coagulase-negative staphylococcus (Infections and infestations) | 1 (1)
Coronavirus NL63 (Infections and infestations) | 1 (1)
Deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1)
Multi-drug resistant Klebsiella bacteremia (Infections and infestations) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Fungal pneumonia (Infections and infestations) | 3 (3)
Fungal sinusitis (Infections and infestations) | 1 (1)
Graft failure (Investigations) | 2 (2)
Human herpesvirus 6 (Infections and infestations) | 1 (1)
Human metapneumovirus (Infections and infestations) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Liver failure (Hepatobiliary disorders) | 2 (2)
Liver graft-versus-host-disease (Immune system disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2)
Hemolytic anemia (Immune system disorders) | 1 (1)
Multisystem organ dysfunction syndrome (Immune system disorders) | 3 (3)
Febrile neutropenia (Infections and infestations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 9 (10)
Respiratory and metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Rhinovirus (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1)
Superior vena cava syndrome (Cardiac disorders) | 1 (1)
Veno-occlusive disease (Hepatobiliary disorders) | 3 (5)
Vancomycin-resistant Enterococcus (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative Haploidentical BMT (N=96)
Acute kidney injury (Renal and urinary disorders) | 8 (8)
BK virus (Infections and infestations) | 6 (6)
Clostridium difficile (Infections and infestations) | 13 (13)
Cytomegalovirus (Infections and infestations) | 14 (19)
Febrile neutropenia (Infections and infestations) | 7 (7)
Mucositis (Skin and subcutaneous tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes